CLINICAL TRIAL: NCT01873404
Title: A Multicenter, Randomized, Double-Blinded, Placebo-Controlled Study Using a Bayesian Adaptive Design to Assess the Efficacy, Safety, Tolerability, and Serum Exposure of Multiple Doses of BG00010 (Neublastin) in Subjects With Painful Lumbar Radiculopathy
Brief Title: BG00010 (Neublastin) Phase 2 Multiple Dose Adaptive Design in Participants With Painful Lumbar Radiculopathy
Acronym: SPRINT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 103NS201
Record Dates: First submitted 2013-05-07; First posted 2013-06-10 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-04

CONDITIONS: Painful Lumbar Radiculopathy; Sciatica; Radiculopathy
MeSH Terms: conditions — Sciatica; Radiculopathy | interventions — ARTN protein, human; Nerve Growth Factor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BG00010 (Experimental): Administered as an IV injection at various dose levels 3 times per week for 1 week
  Interventions: Drug: BG00010
- Placebo (Placebo Comparator): Matched placebo IV injection 3 times per week for 1 week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BG00010 — As specified in the treatment arm
  Other Names: Neublastin
  Arms: BG00010
Drug: Placebo — As specified in the treatment arm
  Arms: Placebo

SUMMARY:
The primary objective of the study is to assess the efficacy of Intravenous (IV) BG00010 (Neublastin) in improving pain in painful lumbar radiculopathy participants when administered 3 times per week for 1 week.

The secondary objectives of this study in this study population are as follows: To explore the duration of the effect of BG00010 in improving pain; To explore the dose response curve on pain reduction; To assess the safety and tolerability of BG00010; To assess the serum exposure to BG00010.

DETAILED DESCRIPTION:
During the study, frequent assessment of allocation probability will be conducted to guide subsequent randomization of participants into dose groups.

ELIGIBILITY:
Key Inclusion Criteria:

* Body weight ≤133 kg.
* Leg pain radiating, diagnosed as being due to painful lumbar radiculopathy or lumbosacral radiculopathy, the diagnosis of which occurred within ≥6 months and ≤5 years of the time of randomization.
* Objective, documented evidence of painful lumbar radiculopathy involvement
* Lower back pain
* Leg pain
* Male and female subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for 3 months after their last dose of study treatment.

Key Exclusion Criteria:

* History of or positive test result at screening for human immunodeficiency virus, or for hepatitis C virus antibody, or current Hepatitis B infection.
* Clinically significant diseases or conditions as determined by the investigator.
* Major surgery within 30 days prior to the Screening Visit or that is scheduled to occur during the study.
* Previous participation in a study with neurotrophic factors (e.g., nerve growth factor).
* Participation in a study with another investigational drug or approved therapy for investigational use within 3 months prior to Day 1.
* Other unspecified reasons that, in the opinion of the Investigator or Biogen Idec Inc. (Biogen Idec), make the subject unsuitable for enrollment

NOTE: Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2013-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the mean 24-hour average general pain intensity (AGPI) score | At the end of treatment period (Day 6-10)

SECONDARY OUTCOMES:
Change from Baseline in the mean 24-hour average back pain intensity (ABPI) score | At the end of the treatment period (day 6-10)
Change from Baseline in the mean 24-hour average leg pain intensity score (ALPI) | At the end of the treatment period (day 6-10)
Change from Baseline in the individual mean 24-hour average general pain intensity (AGPI) | Up to week 5
Change from Baseline in the individual mean 24-hour average back pain intensity (ABPI) | Up to week 5
Change from Baseline in the individual mean 24-hour average leg pain intensity (ALPI) | Up to week 5
Maximum observed serum concentration (Cmax) of BG00010 | Up to Day 5
Number of participants experiencing adverse events (AEs) | Up to week 9
Number of participants experiencing serious adverse events (SAEs) | Up to week 9
Change from Baseline in Incidence of neutralizing antibodies in serum | Up to week 9

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (25):
- United States (25):
  - Research Site, Phoenix, Arizona
  - Research Site, Fresno, California
  - Research Site, Lomita, California
  - Research Site, Long Beach, California
  - Research Site, Pasadena, California
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Orlando, Florida
  - Research Site, Sarasota, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Sunrise, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Columbus, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Bloomington, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Evansville, Indiana
  - Research Site, Overland Park, Kansas
  - Research Site, Brockton, Massachusetts
  - Research Site, Lincoln, Nebraska
  - Research Site, Raleigh, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Duncansville, Pennsylvania
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah